CLINICAL TRIAL: NCT05101564
Title: An Umbrella, Randomized, Controlled, Pre Operative Trial Testing Integrative Subtype Targeted Therapeutics in Estrogen Receptor Positive, HER2-Negative Breast Cancer
Brief Title: Umbrella Trial of Subtype-Targeted Therapies in ER+/HER2- Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Lee Caswell-Jin (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Novartis Pharmaceuticals (Industry); Effector Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Lee Caswell-Jin, Assistant Professor of Medicine (Oncology), Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-52869; NCI-2023-02578 (Other: NCI- Clinical Trials Reporting Program)
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer; ER Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib; Tamoxifen; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (14):
- IC1:Alpelisib in combination with Tamoxifen (closed to enrollment) (Experimental): Integrative subtype IC1, Treatment (14 days, - 2 or + 7 days): Take assigned alpelisib pills, 300 mg (two 150 mg tablets) with food, once daily by mouth. Tamoxifen pills, 20 mg once daily by mouth
  Interventions: Drug: Alpelisib; Drug: Tamoxifen
- IC1:Tamoxifen (closed to enrollment) (Active Comparator): Integrative subtype 1, Treatment (14 days, -2 to +7 days): Take assigned tamoxifen pills, 20 mg once daily by mouth
  Interventions: Drug: Tamoxifen
- IC2:Zotatifin in combination with Fulvestrant (Experimental): Integrative subtype 2, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) should be administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Zotatifin; Drug: Fulvestrant
- IC2:Fulvestrant (Active Comparator): Integrative subtype 2, Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Fulvestrant
- IC3:Zotatifin in combination with Fulvestrant (Experimental): Integrative subtype 3, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) should be administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Zotatifin; Drug: Fulvestrant
- IC3:Fulvestrant (Active Comparator): Integrative subtype 3, Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1. on Day 1.
  Interventions: Drug: Fulvestrant
- IC4:Zotatifin in combination with Fulvestrant (Experimental): Integrative subtype 4, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) should be administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Zotatifin; Drug: Fulvestrant
- IC4:Fulvestrant (Active Comparator): Integrative subtype 4, Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1..
  Interventions: Drug: Fulvestrant
- IC6:Zotatifin in combination with Fulvestrant (Experimental): Integrative subtype 6, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) should be administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Zotatifin; Drug: Fulvestrant
- IC6:Fulvestrant (Active Comparator): Integrative subtype 6, Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Fulvestrant
- IC7:Zotatifin in combination with Fulvestrant (Experimental): Integrative subtype 7, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) should be administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Zotatifin; Drug: Fulvestrant
- IC7:Fulvestrant (Active Comparator): Integrative subtype 7, Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Fulvestrant
- IC8:Zotatifin in combination with Fulvestrant (Experimental): Integrative subtype 8, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) should be administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Zotatifin; Drug: Fulvestrant
- IC8:Fulvestrant (Active Comparator): Integrative subtype 8, Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Alpelisib — Alpelisib 300 mg
  Other Names: Piqray; BYL719
  Arms: IC1:Alpelisib in combination with Tamoxifen (closed to enrollment)
Drug: Tamoxifen — Tamoxifen 20 mg
  Other Names: Soltamox; TAM
  Arms: IC1:Alpelisib in combination with Tamoxifen (closed to enrollment); IC1:Tamoxifen (closed to enrollment)
Drug: Zotatifin — Zotatifin 0.10mg/kg (by weight)
  Other Names: eFT226
  Arms: IC2:Zotatifin in combination with Fulvestrant; IC3:Zotatifin in combination with Fulvestrant; IC4:Zotatifin in combination with Fulvestrant; IC6:Zotatifin in combination with Fulvestrant; IC7:Zotatifin in combination with Fulvestrant; IC8:Zotatifin in combination with Fulvestrant
Drug: Fulvestrant — Fulvestrant 500 mg
  Other Names: Faslodex
  Arms: IC2:Fulvestrant; IC2:Zotatifin in combination with Fulvestrant; IC3:Fulvestrant; IC3:Zotatifin in combination with Fulvestrant; IC4:Fulvestrant; IC4:Zotatifin in combination with Fulvestrant; IC6:Fulvestrant; IC6:Zotatifin in combination with Fulvestrant; IC7:Fulvestrant; IC7:Zotatifin in combination with Fulvestrant; IC8:Fulvestrant; IC8:Zotatifin in combination with Fulvestrant

SUMMARY:
The purpose of this study is to learn if adding a new drug that is targeted at a specific genetic change found in some breast tumors pre-operatively will slow the growth of the tumor more than standard anti-hormone therapy used to treat this type of breast cancer. Different therapies are being tested based on the specific gene changes in the tumor. Not every tumor will have a gene change that is being studied.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the efficacy of investigational agent compared with standard endocrine therapy in in reducing Ki67 values based on digital pathology (QuPath) from baseline to on-treatment biopsy after an specific treatment duration (i.e. 14 days) in ER-positive, HER2-negative tumors (tumor size ≥1 cm) with Ki67 ≥ 10%, for different integrative subtype categories identified at integrative subtype screening.

Secondary Objective: To evaluate the efficacy of investigational agent compared with standard endocrine therapy on the proportion of subjects with Ki67 < 10% after a specific treatment duration (i.e. 14 days)

ELIGIBILITY:
Inclusion Criteria:

* Pre-Screening Phase
* Biopsy-proven ER-positive, HER2-negative breast cancer. ER-positivity and PR-positivity are defined as ≥1% cells staining positive by immunohistochemistry. HER2-negativity is defined by IHC or FISH, per ASCO-CAP 2018 guidelines. Breast tumor must be intact and tumor size must be ≥ 1 cm as measured by ultrasound, mammogram, MRI, or clinical exam. If tumor is locally recurrent, it must be in the breast (not skin, node, or chest wall recurrence). Ki67 may or may not have been done locally but if done locally, must be ≥ 5%. Any nodal status is allowed, as M0 or M1 disease.
* Women or men, age ≥ 18 years old.
* Performance status 0 to 1 (by Eastern Cooperative Oncology Group [ECOG] scale).
* Ability to understand and the willingness to sign a written informed consent document.

Treatment Phase

* Breast tumor classifies as relevant integrative subtype per tumor sequencing performed and analyzed by central laboratory.
* Breast tumor Ki67 score ≥ 10% as assessed by central laboratory.
* Each investigational agent specific inclusion criteria can be found in the agent-specific appendix

Exclusion Criteria:

* Pregnant woman, as confirmed by positive serum hCG test prior to initiating study treatment. Nursing (lactating) woman also not allowed.
* Prior breast cancer-directed therapy (surgery, radiation, chemotherapy, or endocrine therapy) is not allowed, with the exception of people with in-breast recurrences. People with in-breast recurrences cannot have had breast cancer-directed therapy (radiation, chemotherapy, or endocrine therapy; surgery is acceptable) within the 6 months prior to signing the pre-screening consent. Pre-endocrine therapy for breast cancer risk reduction is allowed.
* Known hypersensitivity to study agent (IP) or standard endocrine therapy drug, or to any of the excipients of study agent (IP) or standard endocrine therapy drug.
* Each study agent specific exclusion criteria can be found in the agent-specific appendix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Caswell-Jin, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2: Zotatifin in Combination With Fulvestrant (Treatment Arm): Integrative subtype 2 or 6 Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) was administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant was administered intramuscularly as two 5mL injection on Day 1.
  Zotatifin: Zotatifin 0.10mg/kg (by weight)
  Fulvestrant: Fulvestrant 500 mg
- Cohort 2: Fulvestrant (Control Arm): Integrative subtype 2 or 6, Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant was administered intramuscularly as two 5mL injection on Day 1.
  Fulvestrant: Fulvestrant 500 mg
- Cohort 3:Zotatifin in Combination With Fulvestrant (Treatment Arm): Integrative subtype 3, 4, 7, or 8, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) should be administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant should be administered intramuscularly as two 5mL injection on Day 1.
  Zotatifin: Zotatifin 0.10mg/kg (by weight)
  Fulvestrant: Fulvestrant 500 mg
- Cohort 3:Fulvestrant (Control Arm): Integrative subtype 3, 4, 7, or 8, Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant was administered intramuscularly as two 5mL injection on Day 1. on Day 1.
  Fulvestrant: Fulvestrant 500 mg
Period: Overall Study
Arm/Group | Cohort 2: Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 2: Fulvestrant (Control Arm) | Cohort 3:Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 3:Fulvestrant (Control Arm)
Started | 2 | 2 | 7 | 8
Completed | 2 | 2 | 6 | 8
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2: Zotatifin in Combination With Fulvestrant (Treatment Arm): Integrative subtype 2 or 6, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) was administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant was administered intramuscularly as two 5mL injection on Day 1.
  Zotatifin: Zotatifin 0.10mg/kg (by weight)
  Fulvestrant: Fulvestrant 500 mg
- Cohort 3: Zotatifin in Combination With Fulvestrant (Treatment Arm): Integrative subtype 3, 4, 7, or 8, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) was administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant was administered intramuscularly as two 5mL injection on Day 1.
  Zotatifin: Zotatifin 0.10mg/kg (by weight)
  Fulvestrant: Fulvestrant 500 mg
- Cohort 3: Fulvestrant (Control Arm): Integrative subtype 3, 4, 7, or 8, Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant was administered intramuscularly as two 5mL injection on Day 1. on Day 1.
  Fulvestrant: Fulvestrant 500 mg
- Total: Total of all reporting groups
Arm/Group | Cohort 2: Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 2: Fulvestrant (Control Arm) | Cohort 3: Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 3: Fulvestrant (Control Arm) | Total
Number analyzed (Participants) | 2 | 2 | 7 | 8 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 6 | 4 | 13
  >=65 years | 1 | 0 | 1 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 7 | 8 | 19
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 4 | 2 | 6
  Not Hispanic or Latino | 1 | 2 | 3 | 6 | 12
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 6 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 7 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Ki67
Description: The primary outcome is the percentage change in Ki67 expression comparing pre-treatment to on-treatment specimens. Ki67 values were log-transformed for analysis, and results are summarized as the mean percentage change with 95% confidence intervals.
Time Frame: Measured pre-treatment and after treatment 15 or 19 days, based on the duration specified for the assigned therapy
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Cohort 2: Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 2: Fulvestrant (Control Arm) | Cohort 3: Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 3: Fulvestrant (Control Arm)
Number analyzed (Participants) | 2 | 2 | 6 | 8
percentage | -0.64 [-4.28 to 2.99] | -0.68 [-3.99 to 2.64] | -0.63 [-0.92 to -0.34] | -0.46 [-0.75 to -0.17]

2. Secondary Outcome: Ki67 <10% On-treatment Measurement
Description: The proportions of subjects with Ki67 less than 10% after treatment. The outcome will be reported as a number without dispersion.
Time Frame: 15 or 19 days, based on the duration specified for the assigned therapy
Measure: Number; unit: participants
Groups:
- Cohort 2: Zotatifin in Combination With Fulvestrant (Treatment Arm): Integrative subtype 2 or 6,Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) was administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant was administered intramuscularly as two 5mL injection on Day 1.
  Zotatifin: Zotatifin 0.10mg/kg (by weight)
  Fulvestrant: Fulvestrant 500 mg
Arm/Group | Cohort 2: Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 2: Fulvestrant (Control Arm) | Cohort 3: Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 3: Fulvestrant (Control Arm)
Number analyzed (Participants) | 2 | 2 | 6 | 8
participants | 1 | 1 | 3 | 5

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Cohort 3:Zotatifin in Combination With Fulvestrant (Treatment Arm): Integrative subtype 3, 4, 7, or 8, Treatment (14 days, - 2 to +7 days). Zotatifin (calculated by weight, 0.10 mg/kg) was administered as a 60-minute IV infusion on Days 1. A total of 500 mg Fulvestrant was administered intramuscularly as two 5mL injection on Day 1.
  Zotatifin: Zotatifin 0.10mg/kg (by weight)
  Fulvestrant: Fulvestrant 500 mg
- Cohort 3: Fulvestrant (Control Arm): Integrative subtype 3, 4, 7, or 8,Treatment (14 days, - 2 to +7 days) A total of 500 mg Fulvestrant was administered intramuscularly as two 5mL injection on Day 1. on Day 1.
  Fulvestrant: Fulvestrant 500 mg
Arm/Group | Cohort 2: Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 2: Fulvestrant (Control Arm) | Cohort 3:Zotatifin in Combination With Fulvestrant (Treatment Arm) | Cohort 3: Fulvestrant (Control Arm)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 7/7 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2: Zotatifin in Combination With Fulvestrant (Treatment Arm) (N=2) | Cohort 2: Fulvestrant (Control Arm) (N=2) | Cohort 3:Zotatifin in Combination With Fulvestrant (Treatment Arm) (N=7) | Cohort 3: Fulvestrant (Control Arm) (N=8)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Infections and infestations) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
bruising (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT05101564/Prot_SAP_000.pdf